CLINICAL TRIAL: NCT06675903
Title: Continuous Glucose Monitoring in Kidney Transplant Recipients with Diabetes, Pre-diabetes and Without Diabetes
Brief Title: Continuous Glucose Monitoring (CGM) After Kidney Transplantation
Acronym: CGM-KTx
Status: Recruiting | Type: Observational
Sponsor: Bo Feldt-Rasmussen (Other)
Responsible Party: Sponsor-Investigator, Bo Feldt-Rasmussen, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-24046404
Record Dates: First submitted 2024-10-31; First posted 2024-11-05 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Hyperglycaemia; Kidney Transplantation
Keywords: Kidney transplantation; diabetes; prediabetes; hyperglycaemia; continuous glucose monitoring; CGM
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus; Prediabetic State

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Diabetes: Diabetes group defined as type 2 diabetes, type 1 diabetes, receiving glucose-lowering therapy, FPG ≥ 7 mmol/l, HbA1c ≥ 48mmol/l or non-fasting plasma glucose ≥11.1 mmol/l
- No diabetes: No diabetes defined as HbA1c <42mmol/mol or FPG<6.1 mmol/L
- Prediabetes: Prediabetes group defined as HbA1c 42-47 mmol/mol or FPG 6.1-6.9 mmol/L

SUMMARY:
This study examines glucose levels measured by continuous glucose monitoring (CGM) in the immediate period following kidney transplantation among recipients with diabetes, without diabetes, and with pre-diabetes.

The primary objective is to analyse differences in mean sensor glucose between these three groups.

CGMs are applied to participants within 72 hours after kidney transplantation, with a total of 54 participants divided equally across the three groups (18 in each).

Secondary objectives include assessing additional glucose profile indices, adherence to relevant guidelines, changes in HbA1c, the impact of immunosuppression and steroid dosage, and beta cell function.

DETAILED DESCRIPTION:
Introduction:

Hyperglycaemia is a common medical complication within the first two weeks following kidney transplantation. High doses of prednisone induce a state of insulin resistance, which can cause hyperglycaemia or disrupt glucose regulation in patients with pre-existing diabetes. Current guidelines recommend daily blood glucose monitoring (BGM), defined as four daily glucose measurements during the first four days post-transplant, with insulin administered to maintain stable glucose levels. Minor studies using continuous glucose monitoring (CGM) suggest that patients, particularly those with diabetes, are prone to dysregulation. Early and optimised treatment of post-surgical hyperglycaemia may reduce the risk of later post-transplant diabetes mellitus (PTDM) and associated cardiovascular mortality and loss of graft function.

Objectives:

This study aims to investigate differences in glucose profiles during the initial two weeks following kidney transplantation among patients with diabetes, prediabetes, and no diabetes. We hypothesise that patients with pre-existing diabetes will exhibit the highest glucose levels, despite insulin treatment.

Background:

Patients with end-stage kidney disease require kidney replacement therapy, provided through haemodialysis, peritoneal dialysis, or kidney transplantation. Kidney transplantation is generally considered the best option in terms of quality of life and cost-effectiveness. However, kidney transplant recipients require complex immunosuppressive regimens and present an increased susceptibility to infection, malignancy, cardiovascular disease, and diabetes risk.

Post-transplant hyperglycaemia frequently develops in the early weeks after kidney transplantation. This condition resembles type 2 diabetes and necessitates glucose-lowering therapy to mitigate its harmful effects. Hyperglycaemia primarily arises due to high-dose glucocorticoids or surgical stress, both of which induce insulin resistance. It is characterised by a plasma glucose level of ≥7.0 mmol/L or a 2-hour plasma glucose level of ≥11.1 mmol/L after an oral glucose tolerance test.

Early post-transplant hyperglycaemia exerts stress on pancreatic beta cells, which may contribute to the development of PTDM later on. Although hyperglycaemia may resolve with reduced doses of glucocorticoids and calcineurin inhibitors, kidney transplant recipients remain at an increased risk of PTDM, with an estimated one-year risk of 10-15%. PTDM can be diagnosed three months post-transplant, once patients are on stable immunosuppressive therapy and exhibit stable kidney graft function. Insulin resistance and steroid-induced weight gain play a significant role in the development of PTDM, with hyperglycaemia from steroids often presenting as elevated postprandial glucose levels. Glucose measurement 7-8 hours after prednisolone administration may be optimal for detecting hyperglycaemia, but an oral glucose tolerance test is considered even more effective.

Identifying post-transplant hyperglycaemia early is critical for reducing the risk of developing PTDM. Long-term, PTDM is associated with an increased risk of cardiovascular mortality and reduced graft survival.

Continuous glucose monitoring (CGM) are gradually becoming more widely used for glucose monitoring in patients with impaired glucose levels. Plasma glucose is measured every 5-15 minutes, depending on the model used, usually for 10-14 days. A sensor measures interstitial glucose, which is converted to plasma glucose levels. This provides precise measurements of plasma glucose, including during sleep and periods of variability. This enables clinicians to optimise treatment based on comprehensive glycaemic profiles.

Other metrics, such as time in range and glucose management indicator (GMI) - a calculated estimation of HbA1c based on mean glucose - are also provided by the CGM.

Few studies have explored glucose profiles by CGM immediately after kidney transplantation. A small study found a significant association between mean sensor glucose 3-5 days after renal transplantation and later development of PTDM. Data was based on glucose profiles measured by CGM on 28 kidney transplanted patients and glucose profiles also revealed higher glucose levels in the afternoon and early evening.

Design and Population:

This single-centre observational study will be conducted at Rigshospitalet in Copenhagen, Denmark. A total of 54 participants will be included, divided into three groups based on their diabetes status or most recent fasting plasma glucose and HbA1c measurements before transplantation:

* Diabetes group (n=18)
* No diabetes group (n=18)
* Prediabetes group (n=18)

Methods:

Kidney transplant recipients will receive information about the study prior to or upon admission before transplantation. Patients who meet the inclusion and exclusion criteria and provide written, informed consent will be enrolled in one of the three groups.

A CGM will be applied within 72 hours of kidney transplantation, and additional blood samples (HbA1c, C-peptide, and insulin) will be taken. The CGM will measure glucose levels for 10-14 days, depending on the model used, and additional blood samples will be collected upon CGM removal. Data during the CGM monitoring period, including medication, complications, blood samples, and vital signs, will be obtained from patients' records. Since the CGMs are double-blinded, treating physicians will adhere to guidelines for managing hyperglycaemia.

Statistical Analysis:

We will compare the mean sensor glucose levels across the three groups using analysis of variance (ANOVA) or the Kruskal-Wallis test, depending on data distribution. Post-hoc tests will identify specific group differences in glucose levels. Regression analyses, such as logistic and linear regression, will examine associations between the groups on secondary outcomes, and multivariate analysis will be conducted.

Ethical Considerations:

This study aims to contribute to understanding glucose profiles post-kidney transplantation, ultimately improving monitoring and treatment for post-transplant hyperglycaemia. Informed consent is essential to ensure participants understand the study's purpose and procedures. Special considerations will be taken to protect the autonomy and well-being of kidney transplant recipients, a potentially vulnerable population

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before CGM application
* Male or female; age: ≥18 years
* Kidney transplantation

Exclusion Criteria:

* Unable to cooperate to CGM the first ten days after surgery
* Allergic to plasters in CGM units
* Combined kidney and liver or pancreatic transplantation
* Graft loss/rejection within first 48 hours after transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult kidney transplant recipients at Rigshospitalet, Copenhagen, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Difference in Mean Sensor Glucose | 10 days
  Mean sensor glucose (mmol/L) evaluated by CGM

SECONDARY OUTCOMES:
Time in range (%) | 10 days
  Time within 3.9-10.0 mmol/L as evaluated by CGM
Compliance with applicable guideline (%) | 10 days
  Based on capillary blood glucose (mmol/L) and daily insulin dose (IE per day)
Time in hypoglycaemia (%) | 10 days
  Time in level 1 (3.0-3.8 mmol/L) and level 2 (below 3.0 mmol/L]) evaluated by CGM
Time in tight glycaemic range (%) | 10 days
  Time in 3.9-7.8 mmol/L evaluated by CGM
Time i hyperglycaemia (%) | 10 days
  Time in level 1 (10.1-13.9 mmol/L) and level 2 (above 13.9 mmol/L) evaluated by CGM
Glucose variability | 10 days
  Standard deviation [mmol/L] and coefficient of variation [%]) evaluated by CGM
Glucose management indicator (GMI) (mmol/mol and %) | 10 days
  Evaluated by CGM
Number of hyperglycaemic events (Number/days measured) | 10 days
  Defined as glucose ≥10.0mmol/L for more than 15 minutes measured by CGM
Number of hypoglycaemic events (Number/days measured) | 10 days
  Defined as glucose <3.9mmol/L for more than 15 minutes measured by CGM

OTHER OUTCOMES:
HbA1c | 10 days
  Changes in HbA1c (mmol/mol and %) 10-14 days after kidney transplantation
Daily dose of immunosuppressant | 10 days
  prednisone, tacrolimus, cyclosporine, mycophenolate mofetil
HOMA | 10 days
  HOMA calculated from fasting glucose (mmol/L) and fasting plasma insulin (pmol/L) at time of transplantation and 10-14 days after kidney transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, DK, Denmark

IPD SHARING:
Plan to Share IPD: No